CLINICAL TRIAL: NCT01476761
Title: The Cardica MicroCutter in Surgical Stapling: A Prospective, Open-label, Multi-center Study
Brief Title: MicroCutter in Surgical Stapling - European Trial I
Acronym: MET1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cardica, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 2011-01
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Thoracic
Keywords: Surgical tissue resection; Tissue dissection; Tissue transection; Anastomosis of gastrointestina tissue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MicroCutter Stapling Device (Active Comparator): Patients undergoing surgical treatment with the MicroCutter Stapling Device
  Interventions: Device: Microcutter XPRESS and Microcutter XCHANGE

INTERVENTIONS:
Device: Microcutter XPRESS and Microcutter XCHANGE — Surgical stapling devices
  Other Names: MicroCutter XPRESS30; MicroCutter XPRESS45; MicroCutter XCHANGE30

SUMMARY:
The purpose of this study is to evaluate safety of the Microcutter stapling /cutting device in patients requiring the transection, resection or anastomosis of gastrointestinal tissue in a post-market approval study.

DETAILED DESCRIPTION:
A prospective, open label, multi-center non-inferiority safety study with an all-comers enrollment of patients requiring surgical stapling of the stomach and/or intestine according to the labeled indications contained in the approved labeling. Up to 178 subjects consented for a 1-month clinical follow-up evaluation will be enrolled. Primary endpoint is to statistical non-inferiority of composite major adverse event rate (composite of infection (non-dermal), dehiscence, bleeding, and strictures) in study patients when compared to composite major adverse event rate (composite of infection (non-dermal), dehiscence, bleeding, and strictures) as derived from a comprehensive analysis of the medical literature. The comparison will be performed for cumulative events up to 30 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

- All patients requiring surgical treatment where the use of a surgical stapler is anticipated

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Composite adverse event rate | up to 30 days postoperatively
  Composite event rate is a compilation of the following stapling related adverse event rates: bleeding, leakage, stricture and infection

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kithe, M.D., Principal Investigator — DRK-Krankenhaus Clementinenhaud, Hannover
Locations (1):
- DRK-Krankenahus Clementinenhaus, Hanover, Germany

REFERENCES:
- See also: Manufacturer of MicroCutter — http://www.cardica.com